CLINICAL TRIAL: NCT07122752
Title: Feasibility, Safety and Patient Reported Outcomes of 3D-Printed Externally-applied Cranial Orthosis (PEACO) After Decompression Craniectomy in Clinical Settings: A Retrospective Comparison Study of Monitored Versus Unmonitored Protocols
Brief Title: Feasibility and Outcomes of 3D-printed External Cranial Orthosis After Craniectomy
Status: Active, not recruiting | Type: Observational
Sponsor: Tan Tock Seng Hospital (Other)
Responsible Party: Principal Investigator, Chua Sui Geok, Karen, Senior Consultant Dr (MD), Tan Tock Seng Hospital
Other Study IDs: DSRB 2025/1218
Record Dates: First submitted 2025-07-31; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Traumatic Brain Injury; Acquired Brain Injury; Brain Tumor; Stroke
Keywords: Cranial Orthosis; 3D Printing; Decompression Craniectomy; Retrospective Study; Head Protection Device; Monitored Protocol; Unmonitored Protocol
MeSH Terms: conditions — Brain Injuries, Traumatic; Brain Injuries; Brain Neoplasms; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Version 1 Head protection Device 2021: Version 2 Head protection device 2025

SUMMARY:
This study will compare the outcomes of a current clinical implementation of PEACO designed for one-handed donning and doffing with carer-monitoring with a previous prototype (HPPD) requiring carer-donning and doffing with therapist monitoring.

DETAILED DESCRIPTION:
The study aims to:

1. Evaluate the feasibility, safety and clinical outcomes of a 3D-printed externally applied cranial orthosis (PEACO) in a clinical setting (unmonitored protocol)
2. Comparison of device A - 2021 Head Protection Prototype Device (HPPD) (DSRB 2019/00155)-monitored protocol with device B (PEACO).

ELIGIBILITY:
Inclusion Criteria:

* Unilateral decompressive craniectomy (DC)
* Acute Stroke or traumatic brain injury
* >30 days post DC
* Healed surgical wounds, non-bulging flaps
* Presence of caregiver supervision

Exclusion Criteria:

* Vegetative or minimally responsive state
* Uncontrolled medical illnesses, e.g. sepsis, delirium, active malignancy
* Life expectancy < 6 months
* Unhealed or infected post-DC neurosurgical wounds
* Known allergy to investigational products

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NA as no patient is recruited for this study as the outcomes involve retrospective data as part of a clinical service audit.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2025-07-29 (Actual); Primary Completion 2026-08-29 (Estimated); Study Completion 2026-08-29 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (safety and tolerability) | 30 minutes post fitting (version 1 and 2)
  The therapist will assess patient in terms of pain, redness, skin imprints and pruritus' on patient's skin after wearing the cranial cap. This is to allow the understanding of the incidence of the treatment-emergent adverse events (safety and tolerability).
Patient Reported Outcome Measures (PROMS) PROMs (compliance) | 2023-2025
  The patient will be sent a questionnaire. The question relating to compliance is "Approximately, how many hours of wear per day including rest breaks?" This will allow team to assess feasibility, safety and clinical outcomes.
Patient Reported Outcome Measures (PROMS) PROMs (wearing time) | 2023-2025
  The patient will be sent a questionnaire. The question relating to wearing time is "Approximately, how many hours of wear per day including rest breaks?" This will allow team to assess feasibility, safety and clinical outcomes.
Patient Reported Outcome Measures (PROMS) PROMs (adverse events) | 2023-2025
  The patient will be sent a questionnaire. The question relating to adverse event is "Did you experience any of the following after two hours of wear? This will allow team to assess feasibility, safety and clinical outcomes.
Patient Reported Outcome Measures (PROMS) PROMs (cosmesis rating) | 2023-2025
  The patient will be sent a questionnaire. The question relating to cosmesis rating is "Please rate the appearance of your cranial cap". This will allow team to assess feasibility, safety and clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Karen Chua, MBBS, Principal Investigator — Tan Tock Seng Hospital
Locations (1):
- Tan Tock Seng Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No
no new IP generated

REFERENCES:
- [Background] Chua KSG, Krishnan RR, Yen JM, Plunkett TK, Soh YM, Lim CJ, Chia CM, Looi JC, Ng SG, Rao J. 3D-printed external cranial protection following decompressive craniectomy after brain injury: A pilot feasibility cohort study. PLoS One. 2021 Oct 28;16(10):e0258296. doi: 10.1371/journal.pone.0258296. eCollection 2021. PMID 34710123
- [Background] Fernandez LL, Rodriguez D, Griswold DP, Khun I, Aristizabal S, Aristizabal JH, Richards G, Pavek A, Jayaraman S. Innovative External Cranial Devices for Protecting a Craniectomy Site: A Scoping Review on Noninvasive Approaches for Patients Awaiting Cranioplasty. Neurosurgery. 2025 Apr 1;96(4):713-724. doi: 10.1227/neu.0000000000003157. Epub 2024 Sep 9. PMID 39248525
- [Background] Ma S, Li C, Gu Y, Chen Y, Li X, Wang Q, Xu H. Application of a 3D printed wig protection device after decompressive craniectomy. Sci Rep. 2025 Mar 19;15(1):9545. doi: 10.1038/s41598-025-94246-0. PMID 40108252